CLINICAL TRIAL: NCT02904200
Title: A Randomized Open, Controlled Pilot Investigation Comparing Trauma to the Periwound Skin and Pain During Treatment With Avance NPWT System When Using Two Different Fixations
Brief Title: Clinical Investigation of Two Different Wound Dressings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Avance 02
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-09

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silicon adhesive dressing (Experimental): Sterile soft silicon adhesive dressing
  Interventions: Device: Silicon adhesive dressing
- Acrylic adhesive dressing (Active Comparator): Sterile acrylic adhesive dressing
  Interventions: Device: Acrylic adhesive dressing

INTERVENTIONS:
Device: Silicon adhesive dressing — Sterile soft silicon adhesive dressing
  Arms: Silicon adhesive dressing
Device: Acrylic adhesive dressing — Sterile acrylic adhesive dressing
  Arms: Acrylic adhesive dressing

SUMMARY:
The primary objective of this investigation is to evaluate changes on Peri-Wound skin from baseline to termination when using two different wound dressings

The secondary objectives are to evaluate pain before, during, and after dressing removal from baseline to termination

DETAILED DESCRIPTION:
A prospective randomized clinical investigation will be conducted at two sites in Sweden.

Male or female, 18 years or older with following wound types:

* traumatic, surgical or dehisced wounds,
* venous leg ulcer or pressure ulcer will be included into the clinical investigation.

  32 evaluated subjects (i:e 16 subjects per arm) will be followed during maximum three weeks. The treatment arm (either silicon adhesive dressing or acrylic adhesive dressing). Patients will be randomized using optimal allocation (minimization) balancing for the following baseline variables type of skin (normal/dry/flaky/oily/moist) and age. Eligible patients will be randomized to receive either silicon adhesive dressing or acrylic adhesive dressing in a ratio of 1:1 provided.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic, surgical or dehisced wounds, Venous Leg Ulcer, Diabetic Foot Ulcer or Pressure Ulcer indicated for treatment with NPWT therapy
2. In case of multiple wounds the target wound must be ≥10 cm distant from other wounds. Selection of the target wound is according to the investigator's preference.
3. Peri-wound skin assessable and 5 cm of peri-wound skin present around the wound
4. Male or female, 18 years of age and above
5. Signed Informed Consent

Exclusion Criteria:

1. Dressing sizes does not fit the target wound
2. Unexplored blind tunnels or non-enteric fistula
3. Untreated osteomyelitis
4. Malignant wounds
5. Subjects treated with systemic immunosuppressive or glucocorticosteroids, except subjects taking occasional doses or doses less than 10mg prednisolon/day or equivalent.
6. Wounds with necrotic tissue or eschar (if not adequately debrided)
7. Significantly bleeding wounds, as judged by the investigator
8. Subject not suitable for the investigation according to the investigator's judgment
9. Subject included in other ongoing clinical investigation which could interfere with this investigation, as judged by the investigator
10. Known allergy/hypersensitivity to any of the components included into the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Bergstrom, Principal Investigator — Sundsvalls Sjukhus
Locations (2):
- Sweden (2):
  - Sundsvalls sjukhus, Sundsvall
  - Norrlands Universitetssjukhus, Umeå

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Avance® Film With Safetac®: Sterile soft silicon adhesive dressing
  Silicon adhesive dressing: Sterile soft silicon adhesive dressing
- Avance® Transparent Film: Sterile acrylic adhesive dressing
  Acrylic adhesive dressing: Sterile acrylic adhesive dressing
Period: Overall Study
Arm/Group | Avance® Film With Safetac® | Avance® Transparent Film
Started | 2 (One pat. early terminated on own decision, due to travelling distance between home and hospital.) | 0 (No statistical evaluation was performed because only 2 subjects were included in one arm.)
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The clinical investigation was prematurely closed due to very slow recruitment. Only two subjects were enrolled. Only one went through all visits. No conclusion can be made from the report.
  No statistical evaluation was performed because only 2 subjects were included into the study.
Arm/Group | Avance® Film With Safetac®
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 2
Baseline Pain [Mean (Standard Deviation); unit: score on a scale] — Pain level was obtained at baseline. A visual analog scale (VAS) was used by the subjects to assess pain, with a range from 0 to 100, where 100 indicates the worst possible pain.
  score on a scale | 1.5 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Changes on Peri-Wound Skin
Description: The primary objective of this investigation is to evaluate changes on Peri-Wound skin from baseline to termination when using two different wound dressings. The primary endpoint could not be calculated as intended because the baseline score was not evaluable due to missing values for the one subject that completed follow up. The primary outcome is therefore presented at 12 days. The total of the five scores provide a range from 0 to 15, with higher scores indicating a worse outcome.
  The primary endpoint was assessed through the change in the sum of Peri-Wound Skin outcome scores (0-15) collected at each visit (Visit 1 (baseline), Visit 2 (day 4), Visit 3 (day 7), Visit 4 last visit (day 12)) from baseline to termination. The sum of scores will be obtained from five separate data scores, Redness/Irritation, Flaky, Maceration, Blistering, Skin tears, which will be scored separately with a value between 0 and 3 (None=0, Mild=1, Moderate=2, Severe=3).
Time Frame: Visit 4 last visit (day 12)
Population: No statistical evaluation was performed because only 2 subjects were included into the study and 1 completed follow up (other subject withdrew consent). Due to missing values for the one subject that completed follow up, the primary outcome is presented at 12 days.
Measure: Number; unit: score on a scale
Arm/Group | Avance® Film With Safetac®
Number analyzed (Participants) | 1
score on a scale | 3

2. Secondary Outcome: VAS Scale (0-100mm)
Description: Pain level before, during and after dressing removal. A visual analog scale (VAS) was used by the subjects to assess pain, with a range from 0 to 100, where 100 indicates the worst possible pain.
Time Frame: 0-12 days. Visit 1 (baseline), Visit 2 (day 4), Visit 3 (day 7), Visit 4 last visit (day 12)
Population: No statistical evaluation was performed because only 2 subjects were included into the study and 1 completed follow up (other subject withdrew consent). All data is presented for the one subject throughout their follow up of 4 visits.
Measure: Number; unit: score on a scale (0-100)
Arm/Group | Avance® Film With Safetac®
Number analyzed (Participants) | 1
score on a scale (0-100)
  Visit 1: Pain before application of NPWT | 3
  Visit 2: Pain BEFORE removal of the covering film | 2
  Visit 2: Pain DURING removal of the covering film | 27
  Visit 2: Pain AFTER removal of the covering film | 2
  Visit 2: Pain BEFORE removal of the foam filler | 5
  Visit 2: Pain DURING removal of the foam filler | 2
  Visit 2: Pain AFTER removal of the foam filler | 2
  Visit 3: Pain BEFORE removal of the covering film | 19
  Visit 3: Pain DURING removal of the covering film | 12
  Visit 3: Pain AFTER removal of the covering film | 10
  Visit 3: Pain BEFORE removal of the foam filler | 2
  Visit 3: Pain DURING removal of the foam filler | 5
  Visit 3: Pain AFTER removal of the foam filler | 5
  Visit 4: Pain BEFORE removal of the covering film | 4
  Visit 4: Pain DURING removal of the covering film | 17
  Visit 4: Pain AFTER removal of the covering film | 17
  Visit 4: Pain BEFORE removal of the foam filler | 4
  Visit 4: Pain DURING removal of the foam filler | 6
  Visit 4: Pain AFTER removal of the foam filler | 9

ADVERSE EVENTS:
Time Frame: First Subject In (FSI): 17 Oct 2016 Last Subject Out (LSO): 18 Apr 2017 The subject was followed for 18 days for AE/SAE.
Arm/Group | Avance® Film With Safetac®
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avance® Film With Safetac® (N=2)
Blisters (Skin and subcutaneous tissue disorders) | 1 (1) — One ADE was reported, blister with a probable relationship to the Investigational Product.

LIMITATIONS AND CAVEATS:
Early termination of the study due to slow enrollment. Because baseline score was not evaluable for the one subject that completed follow up, primary outcome is presented at 12 days, and not as intended as the change from baseline to last visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02904200/Prot_SAP_000.pdf